CLINICAL TRIAL: NCT03472521
Title: Prevention of Persistent Pain and Opioid Use in Mothers - POMS
Brief Title: Prevention of Persistent Opioid Use in Mothers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-43964
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Results first posted 2021-11-04 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Opioid Use; Postpartum Disorder; Chronic Pain Syndrome
MeSH Terms: conditions — Puerperal Disorders | interventions — Gabapentin; Exercise

STUDY DESIGN:
Intervention Model Description: Double blind randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A randomization table will be used by the research pharmacy and study drug will be prepared in numbered bottles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gabapentin (Experimental): Gabapentin 300 mg capsules will be prescribed at a starting dose of 1 capsule three times a day and titrated on the recommendation of a chronic pain specialist.
  Interventions: Drug: Gabapentin
- Control (Placebo Comparator): Matched placebo capsules will be prescribed at a starting dose of 1 capsule three times a day and titrated on the recommendation of a chronic pain specialist.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Treatment with analgesic adjutant commonly used for post-operative pain, titrated to effect by chronic pain specialist compared to placebo titration.
  Other Names: Active
  Arms: Gabapentin
Drug: Placebo — Placebo to match gabapentin
  Arms: Control

SUMMARY:
Our previous work has identified the group of women at risk for prolonged pain, opioid use and poor functional recovery after childbirth. The optimal intervention to mitigate this risk is unknown. We propose to test an analgesic adjutant that is commonly used for post-operative pain compared to placebo to improve post-partum recovery.

DETAILED DESCRIPTION:
A small percent of the large population of women who give birth have difficulty with prolonged pain, opioid use and poor functional recovery. This may be the first opiate exposure and significant health challenge in a young woman's life.

In our previous work, we have identified 20% who are at highest risk for prolonged pain and delayed opioid cessation and functional recovery with usual care. Moderate to severe pain on postpartum day 1 is a significant predictor of being in the risk group. The optimal intervention to mitigate this risk is unknown.

We plan to test an intervention of low dose gabapentin or placebo to be escalated by a pain medicine doctor as needed. We hypothesize that additional care of women predicted to be higher need by virtue of their postoperative day one pain score (> 6 x2) despite usual multimodal analgesic care will lead to reduced need for opioid, less pain and more rapid functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* Delivery within 5 days, able to provide informed consent, English speaker

Exclusion Criteria:

* Opiate use disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2021-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Flood, MD, MA, Principal Investigator — Stanford University
Locations (1):
- Lucille Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Komatsu R, Carvalho B, Flood PD. Recovery after Nulliparous Birth: A Detailed Analysis of Pain Analgesia and Recovery of Function. Anesthesiology. 2017 Oct;127(4):684-694. doi: 10.1097/ALN.0000000000001789. PMID 28926443
- [Background] Komatsu R, Carvalho B, Flood P. Prediction of outliers in pain, analgesia requirement, and recovery of function after childbirth: a prospective observational cohort study. Br J Anaesth. 2018 Aug;121(2):417-426. doi: 10.1016/j.bja.2018.04.033. PMID 30032880
- [Derived] Fowler C, Chu AW, Guo N, Ansari JR, Shafer SL, Flood PD. Outpatient Treatment With Gabapentin in Women With Severe Acute Pain After Cesarean Delivery Is Ineffective: A Randomized, Double-Blind, Placebo-Controlled Trial. Anesth Analg. 2023 Jun 1;136(6):1122-1132. doi: 10.1213/ANE.0000000000006429. Epub 2023 Apr 12. PMID 37043404

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin: Gabapentin 300 mg capsules, prescribed at a starting dose of 1 capsule three times a day and titrated on the recommendation of a chronic pain specialist.
- Control: Matched placebo capsules, prescribed at a starting dose of 1 capsule three times a day and titrated on the recommendation of a chronic pain specialist.
Period: Overall Study
Arm/Group | Gabapentin | Control
Started | 41 | 37
Received Allocated Intervention | 41 | 37
Completed | 35 | 34
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 3 | 2
Not completed — Discontinued intervention | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Control | Total
Number analyzed (Participants) | 41 | 37 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 37 | 78
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 37 | 78
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 11 | 25
  Not Hispanic or Latino | 27 | 26 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 0 | 2 | 2
  Asian | 12 | 13 | 25
  Caucasian | 15 | 13 | 28
  Pacific Islander | 1 | 0 | 1
  Other | 10 | 7 | 17
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 37 | 78

OUTCOME MEASURES:

1. Primary Outcome: Time to Opioid Cessation as a Measure of Opioid Utilization
Time Frame: Up to 12 weeks
Population: Participants who completed the protocol are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Gabapentin | Control
Number analyzed (Participants) | 35 | 34
weeks | 2 [1 to 4] | 2 [1 to 3]

2. Secondary Outcome: Pain Report
Description: Number of weeks after delivery until resolution of pain as reported by participants. Pain score was averaged each week from daily reporting by participants using a numerical rating scale (range: 1-10, 1 = no pain; 10 = worst pain).
Time Frame: 12 weeks
Population: Participants who completed the protocol are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Gabapentin | Control
Number analyzed (Participants) | 35 | 34
weeks | 7 [5 to 12] | 12 [6 to 12]

3. Secondary Outcome: Functional Recovery
Description: Functional recovery was assessed as the number of weeks after delivery until participants reported they were able to return to pre-delivery function.
Time Frame: 12 weeks
Population: Participants who completed the protocol are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Gabapentin | Control
Number analyzed (Participants) | 35 | 34
weeks | 8 [5 to 12] | 11 [6 to 12]

4. Other Pre Specified Outcome: Fatigue
Description: PROMIS Fatigue 4 questionnaire will be used to assess fatigue as a modifier of the above outcomes.
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Depression
Description: PROMIS Depression 4 questionnaire will be used to assess fatigue as a modifier of the above outcomes.
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Anxiety
Description: PROMIS Anxiety 4 questionnaire will be used to assess fatigue as a modifier of the above outcomes.
Time Frame: 12 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: PROMIS Physical Function
Description: PROMIS Physical Function questionnaire will be used to assess fatigue as a modifier of the above outcomes.
Time Frame: 12 weeks after delivery
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Steps
Description: Fitness tracker measured steps
Time Frame: 12 weeks after delivery
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Sleep
Description: Fitness tracker measured sleep
Time Frame: 12 weeks after delivery
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Heart Rate
Description: Fitness tracker measured heart rate
Time Frame: 12 weeks after delivery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Gabapentin | Control
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/37
Other Adverse Events (participants affected / at risk) | 0/41 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT03472521/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT03472521/SAP_001.pdf